CLINICAL TRIAL: NCT02828579
Title: The Impact of Bariatric Surgery on Non-alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, MD, PhD, Jagiellonian University
Other Study IDs: JagiellonianU-04
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Obesity; NAFLD
Keywords: obesity; bariatric surgery; non-alcoholic fatty liver disease
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patient with morbid obesity defined as a BMI above 40kg/m2 or 35kg/m2 with comorbidities who are qualified for bariatric surgery.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic Sleeve Gastrectomy (LSG) Laparoscopic Roux-en-Y Gastric Bypass (LRYGB)

SUMMARY:
Up to 300 million people have a BMI over 30kg/m2. Obesity is the cause of many serious diseases, such as type 2 diabetes, hypertension and NAFLD. Bariatric surgery is the only effective method of achieving weight loss in patients with morbid obesity.

The aim of the study is to assess the impact of bariatric surgery on non-alcoholic fatty liver disease in patients operated on due to morbid obesity.

DETAILED DESCRIPTION:
Investigators include 20 patients qualified for the bariatric procedure with BMI > 40 kg/m2 or a BMI > 35kg/m2 with the presence of comorbidities. The average body weight in the group was 143.85kg with an average BMI of 49.16kg/m2. Before the procedure, investigators evaluated the severity of the non-alcoholic fatty liver disease in each patient using the Sherif Saadeh ultrasound scale. Investigators also evaluated the levels of the liver enzymes. Follow up was performed twelve months after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients at the age of 18-60, meeting the criteria of qualification for the surgical treatment of obesity, i.e. BMI > 40 kg/m2 or BMI > 35 kg/m2 together with accompanying diseases.

Exclusion Criteria:

* chronic mental diseases
* addictions
* earlier bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The analysis included prospectively collected data from consecutive patients electively operated for morbid obesity in 2015.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
NAFLD | 12 months
  Ultrasound assessment of the severity of NAFLD with the Sherif-Saadeh scale.

SECONDARY OUTCOMES:
Weight loss after bariatric surgery | 12 months after surgery
  Excess Body Mass Index loss (EBMIL)
Comorbidities | 12 months after surgery
  Number of patients with hypertension and diabetes
Liver function impairment | 12 months after surgery
  Standard set of blood liver enzymes including aspartate aminotransferase (AST) and alanine aminotransferase (ALT)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Major, MD, PhD, Principal Investigator — 2'nd Department of General Surgery, Jagiellonian University Medical College

IPD SHARING:
Plan to Share IPD: No
data not entered

REFERENCES:
- [Result] Pirvulescu I, Gheorghe L, Csiki I, Becheanu G, Dumbrava M, Fica S, Martin S, Sarbu A, Gheorghe C, Diculescu M, Copaescu C. Noninvasive clinical model for the diagnosis of nonalcoholic steatohepatitis in overweight and morbidly obese patients undergoing bariatric surgery. Chirurgia (Bucur). 2012 Nov-Dec;107(6):772-9. PMID 23294957
- [Result] Saadeh S, Younossi ZM, Remer EM, Gramlich T, Ong JP, Hurley M, Mullen KD, Cooper JN, Sheridan MJ. The utility of radiological imaging in nonalcoholic fatty liver disease. Gastroenterology. 2002 Sep;123(3):745-50. doi: 10.1053/gast.2002.35354. PMID 12198701
- [Result] Picot J, Jones J, Colquitt JL, Gospodarevskaya E, Loveman E, Baxter L, Clegg AJ. The clinical effectiveness and cost-effectiveness of bariatric (weight loss) surgery for obesity: a systematic review and economic evaluation. Health Technol Assess. 2009 Sep;13(41):1-190, 215-357, iii-iv. doi: 10.3310/hta13410. PMID 19726018
- [Result] Fan JG, Zhu J, Li XJ, Chen L, Lu YS, Li L, Dai F, Li F, Chen SY. Fatty liver and the metabolic syndrome among Shanghai adults. J Gastroenterol Hepatol. 2005 Dec;20(12):1825-32. doi: 10.1111/j.1440-1746.2005.04058.x. PMID 16336439
- [Result] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166